CLINICAL TRIAL: NCT01178229
Title: AWARNESS THROUGH MOVEMENT PHYSIOTERAPEUTIC TECHNIQUE INCREASED THE AIRWAY DIMENSIONS OF BRUXIST CHILDREN: A SINGLE BLIND RANDOMIZED CLINICAL TRIAL.
Brief Title: Physiotherapy on the Airway of Bruxist Children
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: CES University (Other)
Responsible Party: Claudia Restrepo, Director CES-LPH Research Group. CES University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: via aerea 01
Record Dates: First submitted 2010-08-05; First posted 2010-08-10 (Estimated); Last update posted 2010-08-10 (Estimated); Status verified 2006-07

CONDITIONS: Sleep Bruxism; Airway Remodeling; Physical Therapy Modalities
Keywords: Sleep bruxism; Airway remodeling; Physical therapy modalities; Child preschool.
MeSH Terms: conditions — Sleep Bruxism; Airway Remodeling | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Physiotherapy (Experimental): group of bruxist children that received physiotherapy to change the head posture
  Interventions: Other: Physiotherapy
- Control (No Intervention): Group of bruxist children that did not receive treatment

INTERVENTIONS:
Other: Physiotherapy — The physiotherapeutic intervention was based on the Awareness through Movement technique. Ten sessions were planed. Each session lasted three hours.
  The children of the experimental group and their parents were guided by two physiotherapist and the sessions took place in a room rounded by mirrors.
  Each session developed as follows: presentation to the parents of the somatic awareness technique for each day; movements, games, motor tales and exercises performed by the children; in each session, a guide book with cartoons was given to the children and their parents to reinforce the exercises at home to keep a long-term result.
  All the children assisted together to all the sessions and the instructions and instruments given to the children and their parents were the same for all of them.
  Other Names: Awareness through movement
  Arms: Physiotherapy

SUMMARY:
Objective: to evaluate the effects of physiotherapy on the anteroposterior airway size in a group of bruxist children

Question: Is a physiotherapeutic technique aiming at changing the head posture, effective to increase the anteroposterior dimensions of the upper airway in bruxist children?

Hypothesis: The bruxist children treated with physiotherapy will present higher airway dimensions

Design: randomized clinical trial with allocation and blinding of the examiners.

Participants: 3 to 6 year old children with complete primary dentition, dental and skeletal class I occlusion. The participants were classified as bruxist according to the minimal criteria of the ICSD for bruxism. The children were randomized in an experimental (n=13) and a control (n=13) group.

Intervention: A physiotherapeutic intervention using the Awareness through movement technique was applied to the children of the experimental group once a week, until 10 sessions were completed.

Outcome measures: anteroposterior measurements of the nasopharynx, oropharynx and hypopharynx taken in a lateral cephalogram with standardized techniques.

DETAILED DESCRIPTION:
The physiotherapeutic intervention was based on the Awareness Through Movement (ATM) (Goldman 2003, Malmgren-Olson et al 2001) technique. It is an established method of movement re-education where coordination and posture are significant factors. Its proponents believe more effective and efficient actions can emerge from guided exploration of movement that promotes improved attention and awareness and refines the ability to detect information and make perceptual discriminations.

"Awareness through Movement" (ATM) (Stephens et al 2006) is a process which facilitates the learning of strategies for improving organization and coordination of body movement by developing spatial and kinesthetic awareness of body-segment relationships at rest and during motion, awareness of ease of movement, reducing effort in action, and increasing learning of feeling the muscles longer in action and while breathing .

Ten physiotherapeutic sessions were planed during a ten week period, all of them based in children games. Each session lasted three hours.

The children of the experimental group and their parents were guided by two expert physiotherapist previously standardized and the sessions took place in a room rounded by mirrors, where the children were able to see their own movements. The parents helped their own children during the session and in their home plan indicated weekly.

Each session pursued the following steps:

1. Presentation to the parents of the somatic awareness technique for each day.
2. Movements, games, motor tales and exercises performed by the children, guided by the parents and with the guide of the physiotherapists.
3. In each session, a guide book with cartoons was given to the children and their parents to reinforce the exercises at home to keep a long-term result regarding the body and head posture. The guide book was designed and created by physiotherapists, teachers and advertisers that were not participating in the study.
4. After the first session, a feedback was given before starting the next session, so the exercises at home and the difficulties were reviewed and solved.

All the children assisted together to all the sessions and the instructions and instruments given to the children and their parents were the same for all of them.

Error of method There were not statistically significant differences, regarding the age of the two groups.

Standardizations of the examiners and calibration of all the techniques to evaluate the children regarding the clinical examination and the physiotherapeutic evaluation were made on 12 subjects different from the ones included in the investigation. The Intratester (ICC> 0.9 2-way ANOVA) and intertester error (Kappa > 0.7) were not statistically significant.

A calibration of the x-ray technique and a standardization of the digital tracing of both the cephalogram were also performed. The tracing of the cephalogram was standardized between three investigators with 5 x-rays, scanned and traced two times each by each of three of the investigators. To determine the Intratester and intertester reliability, the intraclass correlation coefficient (ICC > 0.3) and Kappa test were applied.

A lateral cephalogram was taken before and immediately after the 10 session physiotherapeutic intervention for each child with the Natural Head Posture technique, described previously by different authors (Solow and Tallgren 1976). The technique is reproducible (Siersbaek-Nielsen and Solow 1982) and allows the clinician to evaluate the natural position of the cervical vertebras and the inclination of the cervical column and head posture.

Afterwards, the digital record of lateral cephalograms were processed in agree with Sayinsu et al 2006, using a program developed under Matlab 5.3 (MathWorks, Inc., MA. USA). Anteroposterior measurements of the nasopharynx, oropharynx and hypopharynx were taken in a lateral cephalogram with standardized techniques.

The method error ranged from 0.27 to 0.64 degrees and the coefficients of reliability from 0.97 to 1.00

Data analysis The sample size was calculated with a confidence of 95% and a statistical power of 80%. The number of subjects required in each group in order to make the comparisons was 12.

Distributions were tested using the Shapiro-Wilk test. The data were compared using the Mann Whitney and chi square tests. For all tests, significance was set at 5% (p < 0.05). Comparisons among and between groups were performed for all the variables (measurements of the airway) in order to answer the research question.

Results: Statistically significant increases were found for the measurements of the oropharynx (3 mm increase. 95% CI 0.22 to 0.32) and hypopharynx (3 mm increase 95% CI 0.11 to 0.20) for the children that received treatment with physiotherapy.

Conclusion: The physical therapy to change the head posture in bruxist children was useful to increase some of the dimensions of the airway in bruxist children.

ELIGIBILITY:
Inclusion Criteria:

* All the children accomplished the minimal criteria of the International Classification of Sleep Disorders (ICSD) for sleep bruxism.
* High anxiety level according to the Conners' Parents' Rating Scales.
* Three to six year old.

Exclusion Criteria:

* Skeletal malocclusions confirmed with cephalometric x-rays
* Dental malocclusions confirmed with dental casts.
* The reports of respiratory diseases.
* Presence of mouth breathing.
* Functional alterations in the body posture, due to any illness

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2006-01; Primary Completion 2007-06 (Actual); Study Completion 2007-11

PRIMARY OUTCOMES:
ad1 | After 10 sessions of physiotherapy
  ad1: Distance between the posterior nasal spine (PNS) and basion (Ba) along the line which intersects the anterior and posterior pharyngeal wall.
ad2 | After the 10 sessions of physiotherapy
  ad2: Distance between the anterior and posterior pharyngeal wall traced perpendicular to the plane sella (S) Ba plane and passing through PNS.
Angle ad1-ad2 | After 10 sessions of physiotherapy
  Angle ad1-ad2: angle formed by ad1 and ad2.
OAW1 | After 10 sessions of physiotherapy
  OAW1: the distance between the points where the functional occlusal plane intersects the anterior and posterior pharyngeal walls.
OAW2 | After 10 sessions of physiotherapy
  OAW2: the distance between points where a line passing through hyoid (hy) and C2 i intersects the anterior and posterior pharyngeal walls.
OAW3 | After 10 sessions of physiotherapy
  OAW3: the distance between the points where a line passing through hy and C4 i intersects the anterior and posterior pharyngeal walls.
Angle OAW2-OAW3 | After 10 sessions of physiotherapy
  Angle OAW2-OAW3: angle formed by OAW2 and OAW3.
SPPS | After 10 sessions of physiotherapy
  SPPS: anteroposterior dimension of the pharynx measured between the posterior pharyngeal wall and the dorsum of the soft palate on a line parallel to the Frankfort horizontal (FH) plane that runs through the middle of a line from PNS to the distal extreme of the soft palate (P).
IPS | after 10 sessions of physiotherapy
  IPS: anteroposterior dimension of the pharynx measured between the posterior pharyngeal wall and the dorsum of the tongue on a line parallel to the FH plane that runs through C2i

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Restrepo, DDS, Principal Investigator — Director CES-LPH Research Group
Locations (1):
- CES Sabaneta Physiotheray Center, Sabaneta, Antioquia, Colombia